CLINICAL TRIAL: NCT06778434
Title: Acid Sphingomyelinase Inhibition to Mitigate the Environmental Exposure Risks of Ultraviolet Light-Induced Actinic Neoplasia and Squamous Cell Carcinoma in US Veterans
Brief Title: The Effect of Topical Imipramine on Photodynamic Therapy-Mediated Immunosuppression on Forearms or Face on US Veterans
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: ONCE-001-24S; IRB-2024-639 (Other: Wright State University IRB); IRB-2024-674 (Other: Wright State University IRB)
Record Dates: First submitted 2025-01-10; First posted 2025-01-16 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Actinic Keratosis; Imipramine; Photodynamic Therapy
MeSH Terms: conditions — Keratosis, Actinic | interventions — Imipramine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Imipramine and Control Vehicle on Forearms (Experimental): 10% imipramine and control vehicle (1.5 ml each) are applied on designated separate dorsal forearm.
  Interventions: Drug: Imipramine; Other: Control Vehicle
- Imipramine and Control Vehicle on Face (Experimental): 10% imipramine and control vehicle (1.5 ml each) are applied on one side of the face for 1 hour.
  Interventions: Drug: Imipramine; Other: Control Vehicle

INTERVENTIONS:
Drug: Imipramine — 10% imipramine
Other: Control Vehicle — polyethylene glycol: dimethyl sulfoxide Solution

SUMMARY:
The purpose of this study is to test the use of topical imipramine in combination with topical photodynamic therapy's (PDT) effect on the effectiveness and pain immunosuppression following treatment. PDT is a commonly used treatment in dermatology for patients who have many pre-cancers (actinic keratosis or "AK") on their skin. These are both FDA-approved medications, but this study is evaluating their use in combination, which has not been evaluated in the past. The investigators have been doing studies using mice that suggest imipramine might reduce immune system suppression by PDT thus allowing it to work better. Subjects whose provider has decided that they may benefit from PDT to treat their skin due to many AK precancerous lesions will be recruited for this study. Please note that the PDT itself is not experimental, only the imipramine treatment to the skin. There is a separate informed consent for the PDT.

ELIGIBILITY:
Inclusion Criteria:

* Adult Males and Females ages 18 and older who are patients at the Dayton VAMC Dermatology clinics
* Skin type must be "Fair", Fitzpatrick type I or II, due to the presence of actinic damage in this population.
* Subjects must have a VA physician's order to receive PDT treatment on their forearms.
* Willing to participate and understand the informed consent document.
* Willing to avoid excess sun exposure/tanning beds to the area to be treated with PDT.
* Has stable transportation to attend study visits at DVA

Exclusion Criteria:

* Currently taking any tricyclic antidepressants (TCAs)
* Currently taking any selective serotonin reuptake inhibitor (SSRI)
* Has Porphyria
* Large tattoos in areas to be tested
* Pregnancy or nursing
* Taking any oral or topical medications that could interfere with the PDT
* Active rashes in the areas

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2029-03-30 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
(Forearm Arm Only): Difference in areas of Candida antigen skin test results with PDT+ imipramine | 7, 30, 90 days post-PDT treatments
  Size of skin reactions from baseline values will be obtained following PDT + vehicle/imipramine using calipers.
(Forearm Arm Only): Difference in redness of Candida antigen skin test results with PDT+ imipramine | 7, 30, 90 days post-PDT treatments
  Redness of skin reactions from baseline values will be obtained following PDT + vehicle/imipramine using mexameter device and thermal imaging.
Difference in numbers of precancerous AK skin lesions with PDT and imipramine on the face | 6, 12 months post-PDT treatment
  Differences in baseline values of AK will be obtained following PDT + vehicle/imipramine by counting and mapping on each side of face/scalp.

SECONDARY OUTCOMES:
Difference in numbers of precancerous AK skin lesions with PDT and imipramine on the forearms | 6, 12 months post-PDT treatment
  Differences in baseline values of AK will be obtained following PDT + vehicle/imipramine by counting and mapping each forearm/wrist.
(Forearm Arm Only): Difference in gene profile of skin following treatment with PDT + imipramine | 7 days post-PDT treatment
  Differences in transcriptome RNA values from baseline will be obtained following PDT + vehicle/impramine by use of tissue RNA-seq with a commercial dermal transcriptomal patch.
Differences in post-PDT redness with PDT + imipramine | 10 min, 30 min, 24 hours post-PDT treatments
  Differences in redness following PDT + imipramine vs PDT + vehicle from baseline values will be obtained using a mexameter device and thermal imaging on face/forearms.
Differences in post-PDT pain with PDT + imipramine | 10 min, 30 min, 24 hours post-PDT treatments
  Differences in pain following PDT + imipramine vs PDT + vehicle from baseline values will be obtained using a visual analog scale on face/forearms.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Travers, MD, Principal Investigator — Dayton VA Medical Center, Dayton, OH
Locations (1):
- Dayton VA Medical Center, Dayton, OH, Dayton, Ohio, United States

IPD SHARING:
Plan to Share IPD: No